CLINICAL TRIAL: NCT06522607
Title: Three-dimensional Analysis of Palatal Morphology of Hypo-, Hyper-, Normodivergent Growing Subjects With Posterior Cross-bite Treated With Rapid Palatal Expander, a Longitudinal Pilot Study.
Brief Title: 3D Analysis of Palatal Morphology of Growing Patients Treated With Rapid Palatal Expander.
Acronym: 3D_MoPal
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6157
Record Dates: First submitted 2024-05-09; First posted 2024-07-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cross-bite; Malocclusion in Children
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: rapid palatal expander — Clinical evaluation of the patients who will be treated with rapid palatal expander for about 6 month.

SUMMARY:
The aim of the present study is to assess the changes of palatal morphology among growing patients with different vertical facial growth patterns treated with rapid palatal expander.

Thirty-six patients referred to "Policlinico Agostino Gemelli" university hospital will be selected. The eligible criteria are posterior cross-bite, mixed dentition, skeletal Class I relationship and prepubertal stage of cervical vertebral maturation. The patients will be split into three groups according to facial divergency (hyper-, hypo-, normodivergent subjects). For each subject, digital dental casts will be recorded before and after treatment using an intraoral scanner. To evaluate two-dimensional maxillary arch changes, linear measurements will be done. To study comprehensively the palatal shape, a set of 240 landmark and semi-landmarks will be digitized on the palatal vault. Then, Geometric Morphometric Analysis (GMA) will be performed to compare morphological variations of the palate among different vertical facial growth pattern groups.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian origin;
* Mixed dentition stage;
* Angle class I or straight step or mesial step molar relationship in primary dentition;
* Skeletal class I (ANB angle between 0° and 5°);
* Vertical dimension evaluated on lateral cephalograms: SN^GoGn>37°: hyperdivergent, SN^GoGn<27°: hypodivergent, 27°<SN^GoGn>37°: normodivergent;
* Cervical vertebral stage 1 or 2 (CVS methods 1-2);
* Posterior cross-bite including deciduous or permanent teeth;
* Presence of good quality pre-treatment records (history, intraoral and extraoral photographs, oral scan, panoramic radiographs, and lateral cephalometric radiographs with reference ruler);
* Oral scan and photographs available for each subject 6 months after the beginning of the therapy;
* Signing the informed consent form.

Exclusion Criteria:

* Previous orthodontic treatment;
* Tooth agenesis or supernumerary teeth;
* Craniofacial abnormalities;
* Tooth impaction in the maxilla;
* Torus palatinus;
* History of dental trauma (avulsion and alveolar/jaw fracture);
* Refusal to sign consent form.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Skeletal class 1 growing patients affected by cross-bite, coming to UOC Dental Clinic, Fondazione Policlinico Agostino Gemelli IRCCS will be enrolled for this study.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphological changes of the palate | 6 months
  The principal aim of this study is to analyze the morphological changes of the palate in growing subjects with posterior cross-bite after rapid palatal expander therapy.
  The intraoral scans of the maxillary arch will be recorded at T0 (before treatment) and T1 (after treatment). To study comprehensively the palatal shape, 3D Geometric Morphometric Method will be applied.
  Pre- and post-treatment intraoral scans will be digitized using Stratovan Checkpoint Software, placing 240 landmarks. The landmark configurations will be superimposed with Procrustes Superimposition.

SECONDARY OUTCOMES:
Geometric Morphometric Analysis of palatal vault among patients with different facial type | 6 months
  The secondary aim of the present study is to compare three-dimensionally maxillary morphological changes after rapid palatal expander therapy among growing subjects with different facial type (hyperdivergent, hypodivergent, normal), using Geometric Morphometric Method. The facial type of each subject will be evaluated on lateral cephalograms, in particular focusing on the vertical skeletal pattern angle.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Clinica Odontoiatrica, Fondazione Poli.., Roma, Italy